CLINICAL TRIAL: NCT00001519
Title: Oxygen Uptake Kinetics During Recovery From Maximal and Submaximal Exercise
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960098; 96-CC-0098
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: Healthy
Keywords: Exercise; Exercise Intensity; Non-Linear Regression; Oxygen Uptake; Recovery; Subject Comparison; Time Constant; VO2
MeSH Terms: conditions — Motor Activity

SUMMARY:
Measurements of dynamic changes in oxygen uptake (VO2 kinetics) during recovery from exercise may describe regulatory control of oxygen transport and utilization and have greater reliability and less inherent risk than assessment of maximal oxygen uptake (VO2max) in patients for whom exercise is limited by pain, excessive fatigue, dyspnea and motivation. The purpose of this pilot study is to evaluate the effect of exercise intensity on the time constant describing changes in VO2 (tauVO2) during recovery from one minute of constant work rate exercise. Five normal healthy volunteers ages 18 and older will perform a progressive maximal aerobic exercise test, using a cycle ergometer, to determine VO2max and lactate threshold (LT) estimated by gas exchange. Each subject will also complete a series of maximal constant work rate tests and submaximal constant work rate tests at 80% LT and 50% of the difference between LT and VO2max (50% delta). Breath by breath variability and VO2 span will be used to determine the number of constant work rate test repetitions, for each subject for each exercise intensity, needed to establish confidence in tauVO2. A mean response profile of VO2 recovery kinetics for each exercise intensity will be analyzed using non-linear regression to determine tauVO2. To examine the effect of exercise intensity on tauVO2, one way analysis of variance will be used to determine whether differences exist among maximal and submaximal (80% LT and 50% delta) time constants. We hypothesize that there will be no significant differences among time constants for VO2 during recovery from maximal and submaximal constant work rate exercise lasting one minute. The results of this study are expected to provide increased understanding of the measurement of VO2 kinetics during recovery.

DETAILED DESCRIPTION:
Measurements of dynamic changes in oxygen uptake (VO2 kinetics) during recovery from exercise may describe regulatory control of oxygen transport and utilization and have greater reliability and less inherent risk than assessment of maximal oxygen uptake (VO2max) in patients for whom exercise is limited by pain, excessive fatigue, dyspnea and motivation. The purpose of this pilot study is to evaluate the effect of exercise intensity on the time constant describing changes in VO2 (tauVO2) during recovery from one minute of constant work rate exercise. Five normal healthy volunteers ages 18 and older will perform a progressive maximal aerobic exercise test, using a cycle ergometer, to determine VO2max and lactate threshold (LT) estimated by gas exchange. Each subject will also complete a series of maximal constant work rate tests and submaximal constant work rate tests at 80% LT and 50% of the difference between LT and VO2max (50% delta). Breath by breath variability and VO2 span will be used to determine the number of constant work rate test repetitions, for each subject for each exercise intensity, needed to establish confidence in tauVO2. A mean response profile of VO2 recovery kinetics for each exercise intensity will be analyzed using non-linear regression to determine tauVO2. To examine the effect of exercise intensity on tauVO2, one way analysis of variance will be used to determine whether differences exist among maximal and submaximal (80% LT and 50% delta) time constants. We hypothesize that there will be no significant differences among time constants for VO2 during recovery from maximal and submaximal constant work rate exercise lasting one minute. The results of this study are expected to provide increased understanding of the measurement of VO2 kinetics during recovery.

ELIGIBILITY:
Normal healthy subjects ages 18 and older.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 1996-06; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sietsema KE, Cooper DM, Perloff JK, Rosove MH, Child JS, Canobbio MM, Whipp BJ, Wasserman K. Dynamics of oxygen uptake during exercise in adults with cyanotic congenital heart disease. Circulation. 1986 Jun;73(6):1137-44. doi: 10.1161/01.cir.73.6.1137. PMID 3698248
- [Background] Hughson RL. Alterations in the oxygen deficit-oxygen debt relationships with beta-adrenergic receptor blockade in man. J Physiol. 1984 Apr;349:375-87. doi: 10.1113/jphysiol.1984.sp015161. PMID 6429319
- [Background] Powers SK, Dodd S, Beadle RE. Oxygen uptake kinetics in trained athletes differing in VO2max. Eur J Appl Physiol Occup Physiol. 1985;54(3):306-8. doi: 10.1007/BF00426150. PMID 4065115